CLINICAL TRIAL: NCT00370344
Title: An Expertise-based Randomized Controlled Trial Comparing Minilaparotomy Cholecystectomy and Laparoscopic Cholecystectomy
Brief Title: Small-incision Open Cholecystectomy or Laparoscopic Cholecystectomy for Gallbladder Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Norrlandstingens Regionförbund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GANO-05-147M
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Biliary Tract Diseases; Gallbladder Diseases; Cholecystitis; Cholecystolithiasis
Keywords: Gallbladder diseases; gallstones; cholecystectomy; minilaparotomy; laparoscopy
MeSH Terms: conditions — Biliary Tract Diseases; Gallbladder Diseases; Cholecystitis; Cholecystolithiasis; Gallstones | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic cholecystectomy (Active Comparator): Operation by experts in laparoscopy.
  Interventions: Procedure: Laparoscopic cholecystectomy
- Small-incision open cholecystectomy (Active Comparator): Operation by experts in small-incision cholecystectomy.
  Interventions: Procedure: Small-incision open cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Operation by experts in laparoscopy. The operation may be performed as laparoscopic or converted to an open operation.
  Arms: Laparoscopic cholecystectomy
Procedure: Small-incision open cholecystectomy — Operation by experts in small-incision open cholecystectomy.
  Arms: Small-incision open cholecystectomy

SUMMARY:
The trial compares minilaparotomy (small-incision) cholecystectomy with (key-hole) laparoscopic cholecystectomy by randomly allocating patients with gallbladder disease to two groups of surgeons, each group being trained for one of the two methods.

DETAILED DESCRIPTION:
Small-incision open cholecystectomy (minilaparotomy) for gallbladder disease has been proven superior to conventional open cholecystectomy. However, it was rapidly overshadowed by laparoscopic cholecystectomy when the latter method was introduced. Today, some 25% of all gallbladder surgery is done with the conventional open cholecystectomy, often on elderly and frail patients. Previous trials comparing minilaparotomy and laparoscopic cholecystectomy have been hampered by surgeons´ different expertise with the two methods. These studies indicate that operation time is shorter and that health care cost is lower for minilaparotomy compared to laparoscopic cholecystectomy, but hard data are scarce. The objective of the present trial is to randomize eligible patients to two groups of surgeons, well trained in either minilaparotomy cholecystectomy or laparoscopic cholecystectomy. Surgeons in the minilaparotomy group will consider extension of the incision when necessary, and surgeons in the laparoscopic group will aim for laparoscopic cholecystectomy with conversion to open cholecystectomy if this is indicated. The design of the study allows wide inclusion criteria for participants, a cost-utility approach in the analysis, and a high external validity of the conclusions reached.

Comparison: Minilaparotomy cholecystectomy compared to laparoscopic cholecystectomy for gallbladder disease.

ELIGIBILITY:
Inclusion Criteria:

1. Cholecystectomy is considered the best available treatment.
2. The patient understands trial information and is capable of making a decision after having received information.
3. The patient wants to undergo cholecystectomy and accepts participation in the trial.

Exclusion Criteria:

1. Age below 18 years.
2. The patient is unable to understand trial information.
3. Competence for both trial groups are lacking when a patient is randomized.
4. The cholecystectomy is part of a more extensive operation (e.g., pancreaticoduodenectomy).
5. The indication of cholecystectomy is proven or suspected cancer of the gallbladder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2006-09; Primary Completion 2011-04 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life, postoperative pain, and health care costs. | Three, seven, eleven, and 30 postoperative days and one year after the operation.

SECONDARY OUTCOMES:
Compliance to evidence-based recommendations for treatment of gallstone complications, postoperative complications, operation time, hospital time, and sick leave. | Thirty days and one year after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Markku M Haapamäki, MD, PhD, Principal Investigator — Umeå University; Mats Rosenmüller, MD, Principal Investigator — Umeå University
Locations (2):
- Sweden (2):
  - Lycksele Hospital, Lycksele, Västerbotten County
  - Department of Surgery and Perioperative Sciences, Umeå University Hospital, Umeå, Västerbotten County

REFERENCES:
- [Background] Devereaux PJ, Bhandari M, Clarke M, Montori VM, Cook DJ, Yusuf S, Sackett DL, Cina CS, Walter SD, Haynes B, Schunemann HJ, Norman GR, Guyatt GH. Need for expertise based randomised controlled trials. BMJ. 2005 Jan 8;330(7482):88. doi: 10.1136/bmj.330.7482.88. PMID 15637373
- [Background] Harju J, Juvonen P, Eskelinen M, Miettinen P, Paakkonen M. Minilaparotomy cholecystectomy versus laparoscopic cholecystectomy: a randomized study with special reference to obesity. Surg Endosc. 2006 Apr;20(4):583-6. doi: 10.1007/s00464-004-2280-6. Epub 2006 Jan 25. PMID 16437283
- [Background] Keus F, de Jong JA, Gooszen HG, van Laarhoven CJ. Laparoscopic versus open cholecystectomy for patients with symptomatic cholecystolithiasis. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD006231. doi: 10.1002/14651858.CD006231. PMID 17054285
- [Background] Keus F, de Jong JA, Gooszen HG, van Laarhoven CJ. Laparoscopic versus small-incision cholecystectomy for patients with symptomatic cholecystolithiasis. Cochrane Database Syst Rev. 2006 Oct 18;2006(4):CD006229. doi: 10.1002/14651858.CD006229. PMID 17054284
- [Derived] Rosenmuller MH, Nilsson E, Lindberg F, Aberg SO, Haapamaki MM. Costs and quality of life of small-incision open cholecystectomy and laparoscopic cholecystectomy - an expertise-based randomised controlled trial. BMC Gastroenterol. 2017 Apr 8;17(1):48. doi: 10.1186/s12876-017-0601-1. PMID 28388942
- [Derived] Rosenmuller MH, Thoren Ornberg M, Myrnas T, Lundberg O, Nilsson E, Haapamaki MM. Expertise-based randomized clinical trial of laparoscopic versus small-incision open cholecystectomy. Br J Surg. 2013 Jun;100(7):886-94. doi: 10.1002/bjs.9133. PMID 23640665